CLINICAL TRIAL: NCT04446429
Title: Anti-Androgen Treatment for COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-DRUG-SARS-004
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; SARS-CoV2; Androgenetic Alopecia; Prostate Cancer; Benign Prostatic Hyperplasia; SARS (Severe Acute Respiratory Syndrome)
Keywords: Anti-Androgen; Proxalutamide
MeSH Terms: conditions — COVID-19; Alopecia; Prostatic Neoplasms; Prostatic Hyperplasia; Severe Acute Respiratory Syndrome | interventions — proxalutamide; Standard of Care

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective, interventional, placebo controlled, double-blinded, randomized parallel assignment study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (Active Comparator): Usual care as determined by the PI
  Interventions: Other: Standard of Care
- Proxalutamide + Usual Care (Experimental): Proxalutamide + Usual care as determined by the PI
  Interventions: Drug: Proxalutamide

INTERVENTIONS:
Drug: Proxalutamide — 200 mg q.d.
  Arms: Proxalutamide + Usual Care
Other: Standard of Care — Standard of care as determined by the PI
  Arms: Usual Care

SUMMARY:
This study is intended to explore the possible protective role of anti-androgens in SARS-CoV-2 infection

DETAILED DESCRIPTION:
During the continuing SARS-CoV-2 (COVID-19) pandemic, several studies have reported a significant difference in the rate of severe cases between adult females and adult males (42% vs 58%).Among children under the age of 14, the rate of severe cases was reported to be extremely low. To explain this difference, several theories have been proposed including cigarette smoking and lifestyle habits. However, no theory fits both the gender difference in severe cases as well as reduced risk in pre-pubescent children. Our past research on male androgenetic alopecia (AGA) has led us to investigate an association between androgens and COVID-19 pathogenesis. In normal subjects, androgen expression demonstrates significant variation between men and women as well as between adults and pre-pubescent children.

SARS-CoV-2 primarily infects type II pneumocytes in the human lung. SARS-CoV-2 enters pneumocytes, by anchoring to the ACE2 cell surface receptor. Prior to receptor binding, viral spike proteins undergo proteolytic priming by the transmembrane protease, serine 2 (TMPRSS2). TMPRSS2 inhibition or knock down reduces ability of SARS-CoV-1 (a related virus to SARS-CoV-2) to infect cells in vitro. Additionally, TMPRSS2 also facilitates entry of influenza A and influenza B into primary human airway cells and type II pneumocytes.

The human TMPRSS2 gene has a 15 bp androgen response element and in humans, androgens are the only known transcription promoters for the TMPRSS2 gene. In a study of androgen-stimulated prostate cancer cells (LNCaP), TMPRSS2 mRNA expression increase was mediated by the androgen receptor. Further, the ACE2 receptor, also critical for SARS-CoV-2 viral infectivity, is affected by male sex hormones with higher activity found in males.

Androgenetic alopecia (AGA), often referred to as male pattern hair loss, is the most common form of hair loss among men. The development of androgenetic alopecia is androgen mediated and is dependent on genetic variants found in the androgen receptor gene located on the X chromosome; thus, it is hypothesized that men with AGA would be more prone to severe COVID-19 disease. The investigators conducted a preliminary observational study of hospitalized COVID-19 patients at two Spanish tertiary hospitals between March 23-April 6, 2020 to test this theory. In total, 41 Caucasian males admitted to the hospitals with a diagnosis of bilateral SARS-CoV-2 pneumonia were analyzed. The mean age of patients was 58 years (range 23-79). Among them, 29 (71%) were diagnosed with AGA (16 (39%) were classified as severe AGA (Hamilton IV or above)) and 12 (29%) did not present clinical signs of AGA. The diagnosis of AGA was performed clinically by a dermatologist. The precise prevalence of AGA among otherwise healthy Spanish Caucasian males is unknown; however, based on published literature, the expected prevalence of a similar age-matched Caucasian population is approximately 31-53%.

Based on the scientific rationale combined with this preliminary observation, the investigators propose to test an anti-androgen as a treatment for patients recently diagnosed with COVID-19.

We have chosen the use of the novel second generation androgen receptor (AR) antagonist proxalutamide as a means for rapid reduction in AR activity. Proxalutamide (GT0918) demonstrates a dual mechanism of action. It is highly effective in inhibiting AR as well as exhibiting pharmacological effects of inducing the down-regulation of AR expression; the mechanism that is not present in bicalutamide and enzalutamide. Additionally, it has been reported that Proxalutamide lowers the expression of ACE2. Both would be beneficial for preventing SARS-CoV-2 entry into lung cells.

This study is intended to explore the possible protective role of anti-androgens in SARS-CoV-2 infection. Provided anti-androgens are effective in reducing the rate of COVID-19 hospitalization, subjects enrolled in this study may experience a lower rate of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

1. Male age ≥18 years old
2. Laboratory confirmed positive SARS-CoV-2 rtPCR test within 7 days prior to randomization
3. Clinical status on the COVID-19 8-point Ordinal Scale of 1 or 2
4. Coagulation: INR ≤ 1.5×ULN, and APTT ≤ 1.5×ULN
5. Subject (or legally authorized representative) gives written informed consent prior to any study screening procedures
6. Subject (or legally authorized representative) agree that subject will not participate in another COVID-19 trial while participating in this study

Exclusion Criteria:

1. Subject enrolled in a study to investigate a treatment for COVID-19
2. Subject taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc…
3. Patients who are allergic to the investigational product or similar drugs (or any excipients);
4. Subjects who have malignant tumors in the past 5 years, with the exception of completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type
5. Subjects with known serious cardiovascular diseases, congenital long QT syndrome, torsade de pointes, myocardial infarction in the past 6 months, or arterial thrombosis, or unstable angina pectoris, or congestive heart failure which is classified as New York Heart Association (NYHA) class 3 or higher, or left ventricular ejection fraction (LVEF) < 50%, QTcF > 450 ms
6. Subjects with uncontrolled medical conditions that could compromise participation in the study(e.g. uncontrolled hypertension, hypothyroidism, diabetes mellitus)
7. Known diagnosis of human immunodeficiency virus(HIV) , hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory）
8. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
9. Estimated glomerular filtration rate (eGFR) < 30 ml/min
10. Severe kidney disease requiring dialysis
11. Subject unlikely to return for day 15 site visit for reasons other then remission
12. Subject (or legally authorized representative) not willing or unable to provide informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 268 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Flavio A Cadegiani, MD, Principal Investigator — Corpometria Institute; Andy Goren, MD, Study Director — Applied Biology, Inc.
Locations (1):
- Corpometria Institute, Brasília, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goren A, McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Dhurat R, Washenik K, Lotti T. What does androgenetic alopecia have to do with COVID-19? An insight into a potential new therapy. Dermatol Ther. 2020 Jul;33(4):e13365. doi: 10.1111/dth.13365. Epub 2020 Apr 8. No abstract available. PMID 32237190
- [Background] Goren A, Vano-Galvan S, Wambier CG, McCoy J, Gomez-Zubiaur A, Moreno-Arrones OM, Shapiro J, Sinclair RD, Gold MH, Kovacevic M, Mesinkovska NA, Goldust M, Washenik K. A preliminary observation: Male pattern hair loss among hospitalized COVID-19 patients in Spain - A potential clue to the role of androgens in COVID-19 severity. J Cosmet Dermatol. 2020 Jul;19(7):1545-1547. doi: 10.1111/jocd.13443. Epub 2020 Apr 23. PMID 32301221
- [Background] McCoy J, Wambier CG, Vano-Galvan S, Shapiro J, Sinclair R, Ramos PM, Washenik K, Andrade M, Herrera S, Goren A. Racial variations in COVID-19 deaths may be due to androgen receptor genetic variants associated with prostate cancer and androgenetic alopecia. Are anti-androgens a potential treatment for COVID-19? J Cosmet Dermatol. 2020 Jul;19(7):1542-1543. doi: 10.1111/jocd.13455. Epub 2020 Jun 14. No abstract available. PMID 32333494
- [Background] Wambier CG, Goren A, Vano-Galvan S, Ramos PM, Ossimetha A, Nau G, Herrera S, McCoy J. Androgen sensitivity gateway to COVID-19 disease severity. Drug Dev Res. 2020 Nov;81(7):771-776. doi: 10.1002/ddr.21688. Epub 2020 May 15. PMID 32412125
- [Background] Wambier CG, Vano-Galvan S, McCoy J, Gomez-Zubiaur A, Herrera S, Hermosa-Gelbard A, Moreno-Arrones OM, Jimenez-Gomez N, Gonzalez-Cantero A, Fonda-Pascual P, Segurado-Miravalles G, Shapiro J, Perez-Garcia B, Goren A. Androgenetic alopecia present in the majority of patients hospitalized with COVID-19: The "Gabrin sign". J Am Acad Dermatol. 2020 Aug;83(2):680-682. doi: 10.1016/j.jaad.2020.05.079. Epub 2020 May 22. PMID 32446821
- [Background] Montopoli M, Zumerle S, Vettor R, Rugge M, Zorzi M, Catapano CV, Carbone GM, Cavalli A, Pagano F, Ragazzi E, Prayer-Galetti T, Alimonti A. Androgen-deprivation therapies for prostate cancer and risk of infection by SARS-CoV-2: a population-based study (N = 4532). Ann Oncol. 2020 Aug;31(8):1040-1045. doi: 10.1016/j.annonc.2020.04.479. Epub 2020 May 6. PMID 32387456
- [Derived] McCoy J, Goren A, Cadegiani FA, Vano-Galvan S, Kovacevic M, Situm M, Shapiro J, Sinclair R, Tosti A, Stanimirovic A, Fonseca D, Dorner E, Onety DC, Zimerman RA, Wambier CG. Proxalutamide Reduces the Rate of Hospitalization for COVID-19 Male Outpatients: A Randomized Double-Blinded Placebo-Controlled Trial. Front Med (Lausanne). 2021 Jul 19;8:668698. doi: 10.3389/fmed.2021.668698. eCollection 2021. PMID 34350193 (Retraction: PMID 35755027 Front Med (Lausanne). 2022 Jun 10;9:964099)

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care: Usual care as determined by the PI
  Usualf Care: Care as determined by the PI
Period: Overall Study
Arm/Group | Usual Care | Proxalutamide + Usual Care
Started | 134 | 134
Completed | 128 (In placebo group, 6 patients were lost to follow-up but were included in intention-to-treat analysis.) | 134
Not Completed | 6 | 0
Not completed — Lost to Follow-up | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Usual Care: Usual care as determined by the PI
  Usual Care: Care as determined by the PI
- Total: Total of all reporting groups
Arm/Group | Usual Care | Proxalutamide + Usual Care | Total
Number analyzed (Participants) | 134 | 134 | 268
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (10.8) | 44.2 (14) | 44.5 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 134 | 134 | 268
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mixed ethnicity (Brazil) | 134 | 134 | 268
Region of Enrollment [Number; unit: participants]
  Brazil | 134 | 134 | 268
Coexisting conditions [Count of Participants; unit: Participants] — At least one coexisting conditions: Type 2 diabetes, Hypertension, COPD and Obesity
  Participants | 20 | 29 | 49

OUTCOME MEASURES:

1. Primary Outcome: COVID-19 Hospitalization
Description: Percentage of subjects hospitalized due to COVID-19
Time Frame: 30 days
Population: All randomized patients were included. 6 patients from the placebo arm lost to follow-up were assumed to be non-hospitalized (COVID-19 8-point ordinal scale 1) and were included in the intention-to-treat analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Care | Proxalutamide + Usual Care
Number analyzed (Participants) | 134 | 134
Participants | 35 | 3

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Usual Care | Proxalutamide + Usual Care
All-Cause Mortality (participants affected / at risk) | 2/134 | 0/134
Serious Adverse Events (participants affected / at risk) | 35/134 | 3/134
Other Adverse Events (participants affected / at risk) | 78/134 | 45/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=134) | Proxalutamide + Usual Care (N=134)
Death (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hospitalization (Respiratory, thoracic and mediastinal disorders) | 35 (35) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Usual Care (N=134) | Proxalutamide + Usual Care (N=134)
Diarrhea (Gastrointestinal disorders) | 20 | 39
Nausea (Gastrointestinal disorders) | 15 | 21
Abdominal pain or discomfort (Gastrointestinal disorders) | 18 | 22
Dyspepsia or Heartburn (Gastrointestinal disorders) | 6 | 23
Fatigue (General disorders) | 71 | 1
Fever (General disorders) | 34 | 2
Disease progression (General disorders) | 43 | 4
Tachycardia (Cardiac disorders) | 45 | 6
Ageusia (Nervous system disorders) | 23 | 13
Anosmia (Nervous system disorders) | 26 | 14
Headache (Nervous system disorders) | 12 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 36 | 16
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 40 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (English Translation) (2020-09-17): https://cdn.clinicaltrials.gov/large-docs/29/NCT04446429/Prot_SAP_001.pdf